CLINICAL TRIAL: NCT02178748
Title: A Phase II Open Label Trial to Investigate the Effect of Schistosoma Mansoni (Sm) Infection on the Immunogenicity of a Candidate TB Vaccine, MVA85A, in BCG-vaccinated African Adolescents
Brief Title: Trial to Investigate the Effect of Schistosoma Mansoni Infection on the Response to Vaccination With MVA85A in BCG-vaccinated African Adolescents
Acronym: TB036
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB036
Record Dates: First submitted 2014-06-03; First posted 2014-07-01 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Phase II; MVA85A; Schistosoma mansoni
MeSH Terms: conditions — Tuberculosis; Schistosomiasis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 (Schistosoma mansoni uninfected): 12-24 BCG-vaccinated volunteers with no helminth infection. Single dose of 1x10^8pfu MVA85A intramuscular vaccination at D0.
  Interventions: Biological: MVA85A
- Group 2 (Experimental): Group 2 (Schistosoma mansoni infected): 12-24 BCG-vaccinated volunteers with helminth infection. Single dose of 1x10^8pfu MVA85A intramuscular vaccination at D0.
  Interventions: Biological: MVA85A

INTERVENTIONS:
Biological: MVA85A — Single dose of 1x10^8pfu MVA85A intramuscular vaccination
  Other Names: Modified Vaccinia Ankara 85A; AERAS-485

SUMMARY:
Mycobacterium tuberculosis (M. tb) is a pathogen with worldwide distribution which infects humans causing tuberculosis (TB), a transmissible disease resulting in very high mortality and morbidity; development of an effective vaccine is a global health priority.

Over a billion people worldwide are infected with one or more helminths. Helminths are parasitic worms, of which Schistosoma mansoni is one species. There is some evidence that helminth infection may affect a person's response to a vaccine. In this trial the investigators hope to investigate whether Schistosoma mansoni infection affects adolescents' responses to a candidate TB vaccine called MVA85A, as adolescents are a crucial target group for an effective TB vaccine.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to enter the trial:

* Healthy adolescents aged 12-17 years (both male and female)
* Resident in the study area for the duration of the study period
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected study vaccination date (by visible BCG scar on examination or written documentation)
* No relevant findings in medical history or on physical examination
* Written informed consent by parent or guardian
* Written informed assent by subject
* Refrain from blood donation during the trial
* Agree to avoid pregnancy for the duration of the trial (female only)
* Able and willing (in the Investigator's opinion) to comply with all the study requirements
* Stool sample negative for S. mansoni (group 1) or positive for S. mansoni infection (group 2), based on the results of the Kato Katz stool analysis
* Willing to delay treatment for schistosomiasis for at least one month (group 2)

Exclusion Criteria

Participants may not enter the trial if ANY of the following apply:

* Clinical, radiological, or laboratory evidence of current active TB disease
* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Previous treatment for active or latent tuberculosis infection
* Shared a residence within one year prior to day 0 with an individual on anti-tuberculosis treatment or with culture or smear-positive pulmonary tuberculosis
* Received a TST within 90 days prior to day 0
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness, drug or alcohol abuse
* History of serious psychiatric condition or disorder
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents within 2 months prior to enrolment
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study vaccine, including eggs
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study
* Positive HBsAg, HCV or HIV antibodies
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the study vaccine for 30 days prior to dosing with the study vaccine, or planned use during the study period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Female currently lactating, confirmed pregnancy or intention to become pregnant during the trial period
* Screening blood sample positive for malaria or Mansonella perstans by microscopy
* Schistosoma mansoni infection intensity greater than 2000 eggs per gram of stool
* Any of the three screening stool samples positive for any helminths on Kato Katz examinations or for S. mansoni or Strongyloides stercoralis by PCR (group 1); or any of the three screening stool samples positive for helminths other than S. mansoni on Kato Katz examinations or for Strongyloides stercoralis by PCR (group 2)
* Screening urine sample positive for S. mansoni infection (group 1)
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
T cell immunogenicity by gamma-interferon ELISPOT of Ag85A response. | 8 weeks
  To compare T cell immunogenicity in adolescents with and without S. mansoni infection.

SECONDARY OUTCOMES:
Evaluation of cytokines in supernatant of stimulated cells using Luminex and flow cytometry of Ag85A response. | 8 weeks
  Effects of S. mansoni infection on other aspects of the immune response following MVA85A immunisation.

OTHER OUTCOMES:
Actively and passively collected data on adverse events. | 8 weeks
  To assess the safety of MVA85A vaccination in BCG-vaccinated African adolescents aged 12-17 years.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Study Director — University of Oxford; Alison Elliot, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- MRC/UVRI Uganda Research Unit on AIDS, Entebbe, Uganda

REFERENCES:
- [Derived] Wajja A, Namutebi M, Apule B, Oduru G, Kiwanuka S, Akello M, Nassanga B, Kabagenyi J, Mpiima J, Vermaak S, Lawrie A, Satti I, Verweij J, Cose S, Levin J, Kaleebu P, Tukahebwa E, McShane H, Elliott AM. Lessons from the first clinical trial of a non-licensed vaccine among Ugandan adolescents: a phase II field trial of the tuberculosis candidate vaccine, MVA85A. Wellcome Open Res. 2018 Sep 19;3:121. doi: 10.12688/wellcomeopenres.14736.1. eCollection 2018. PMID 30687792
- [Derived] Wajja A, Kizito D, Nassanga B, Nalwoga A, Kabagenyi J, Kimuda S, Galiwango R, Mutonyi G, Vermaak S, Satti I, Verweij J, Tukahebwa E, Cose S, Levin J, Kaleebu P, Elliott AM, McShane H. The effect of current Schistosoma mansoni infection on the immunogenicity of a candidate TB vaccine, MVA85A, in BCG-vaccinated adolescents: An open-label trial. PLoS Negl Trop Dis. 2017 May 4;11(5):e0005440. doi: 10.1371/journal.pntd.0005440. eCollection 2017 May. PMID 28472067